CLINICAL TRIAL: NCT00678548
Title: Effect of Positive Guided Imagery on Patients With in or Below-level Chronic Pain Related to Spinal Cord Injury
Brief Title: Effect of Guided Imagery on Patients With Chronic Pain Related to Spinal Cord Injury
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to other projects priority
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4.2007.1943
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- guided imagery (Experimental): CD
  Interventions: Behavioral: Pleasant guided imagery
- pain diary (Active Comparator): Pain diary
  Interventions: Behavioral: Pain diary

INTERVENTIONS:
Behavioral: Pleasant guided imagery — CD with pleasant guided imagery
  Arms: guided imagery
Behavioral: Pain diary — Filling out a pain diary
  Arms: pain diary

SUMMARY:
Chronic pain after spinal cord injury in or below the level of injury is a common problem and can be severe.

The purpose of our study is to investigate the effect of pleasant guided imagery on spinal cord injured patients with chronic pain in or below the level of injury.

DETAILED DESCRIPTION:
The study is a controlled simple blind randomized prospective study. Subjects who live in Trøndelag ( Norway) and who have a traumatic or non traumatic spinal cord injury with chronic pain in or below the level of injury will be included in the study.

Assessments: Pain will be measured with NRS(numeric pain rating scale) and BPIQ (Brief pain intervention questionnaire), anxiety and depression with BDI and BAI (Beck's depression and anxiety inventory) and quality of live with SF36 health survey.

The subjects will be randomized in a treatment and control group. One group will use daily for four weeks a CD with a pleasant guided imagery, the other group will write a short pain diary.

The NRS will be registered daily and the other assessments before and after the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic and non traumatic SCI (spinal cord injury) persons in Trøndelag (Norway)

Exclusion Criteria:

* Not sufficient knowledge of the Norwegian language, cancer, serious cognitive impairment, abuse or dependence of alcohol, narcotics or analgesics and dissociative disorder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Pain intensity | four weeks
  as measured by a numerical rating scale (daily) and Brief pain questionnaire (BPI) (baseline and after 4 weeks)

SECONDARY OUTCOMES:
BDI, BAI and SF36 | pre and postintervention

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Leivseth, Professor MD, Principal Investigator — Norwegian University of Science and Technology